CLINICAL TRIAL: NCT04089865
Title: Blood Loss in Arthroplasty With Oral Versus IV Tranexamic Acid
Brief Title: Oral Versus Intravenous Tranexamic Acid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0882
Record Dates: First submitted 2019-09-06; First posted 2019-09-13 (Actual); Results first posted 2023-06-01 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Blood Loss; Blood Transfusion
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral Tranexamic Acid (TXA) (Experimental): 100 Total Hip Arthroplasty (THA) and 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1950 mg of oral TXA in the pre-operative area.
  Interventions: Drug: Tranexamic Acid
- Intravenous (IV) Tranexamic Acid (TXA) (Active Comparator): 100 Total Hip Arthroplasty (THA) and 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1 g of intravenous (IV) TXA upon transfer to the operating room.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
  Other Names: Lysteda

SUMMARY:
The goal of this randomized clinical control trial is to determine whether oral TXA dosing in THA/TKA result in more blood loss and more transfusions compared to IV TXA dosing in patients undergoing THA/TKA under neuraxial anesthesia. The main questions it aims to answer are:

Does oral TXA dosing in THA/TKA result in more blood loss compared to IV TXA dosing?

Does oral TXA dosing in THA/TKA result in more transfusions compared to IV TXA dosing?

Participants will be randomly assigned to either get the Oral TXA (1950mg) or the IV TXA (1g) on their day of surgery. Researchers will compare these groups to see if any differences emerged. 200 THA patients (100 Oral, 100 IV), 200 TKA patients (100 oral, 100 IV).

DETAILED DESCRIPTION:
Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. The use of TXA in total hip arthroplasty (THA) and total knee arthroplasty (TKA) has resulted in dramatic decreases in operative blood loss and transfusion rates, revolutionizing the field of arthroplasty. The use of TXA, now common, has made autologous blood donation programs largely obsolete. Additionally, it has made perioperative blood transfusion uncommon.

While AAOS guidelines suggest that all three available preparations of TXA (oral, IV, topical) are effective, preferred route of dosing varies by provider and institution. These preferences are based on habit, understanding of pharmacodynamics, and logistical issues regarding effective dosing. Oral TXA is the cheapest option, but some surgeons prefer IV dosing due to concerns regarding efficacy and controlled dosing.

In this study, we seek to compare the efficacy of a single pre-op oral dose of TXA to a single pre-op IV dose of TXA.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip arthroplasty (THA) through a posterior approach
* Patients undergoing total knee arthroplasty (TKA)
* Patients between 18-80 years of age

Exclusion Criteria:

* Patients with >80 years of age
* Patients with a BMI over 40
* Patients undergoing general anesthesia
* Patients with a history of major ipsilateral joint surgery
* Patients on pre-operative anticoagulation or anti-platelet drugs (other than aspirin)
* Patients with a history of bleeding disorders
* Patients with platelets less than 100/nl
* Patients with new-onset/active atrial fibrillation
* Patients with a history of myocardial infarction in the past year
* Patients with a history of a stroke in the past year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Memtsoudis, MD PhD, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Certain individual participant data will be available. Individual participant data that underlie the results reported in a future article, after deidentification (text, tables, figures, appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal, in order to achieve aims in the approved proposal.

RESULTS

PARTICIPANT FLOW:
Groups:
- Total Hip Arthroplasty - Oral TXA: 100 Total Hip Arthroplasty (THA) patients will be randomized to receive 1950 mg of oral TXA in the pre-operative area.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Total Hip Arthroplasty - Intravenous TXA: 100 Total Hip Arthroplasty (THA) patients will be randomized to receive 1 g of intravenous (IV) TXA upon transfer to the operating room.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Total Knee Arthroplasty - Oral TXA: 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1950 mg of oral TXA in the pre-operative area.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Total Knee Arthroplasty - Intravenous TXA: 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1 g of intravenous (IV) TXA upon transfer to the operating room.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
Period: Overall Study
Arm/Group | Total Hip Arthroplasty - Oral TXA | Total Hip Arthroplasty - Intravenous TXA | Total Knee Arthroplasty - Oral TXA | Total Knee Arthroplasty - Intravenous TXA
Started | 100 | 100 | 100 | 100
Completed | 98 | 98 | 93 | 98
Not Completed | 2 | 2 | 7 | 2
Not completed — Withdrawal by Subject | 2 | 2 | 7 | 2

BASELINE CHARACTERISTICS:
Population: Oral Tranexamic Acid (TXA) - 9 subjects did not receive allocated intervention because withdrew from study after allocation/randomization IV Tranexamic Acid (TXA) - 4 subjects did not receive allocated intervention because withdrew from study after allocation/randomization
Groups:
- Total Hip Arthroplasty - Intravenous TXA: 100 Total Hip Arthroplasty (THA) and 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1 g of intravenous (IV) TXA upon transfer to the operating room.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Total: Total of all reporting groups
Arm/Group | Total Hip Arthroplasty - Oral TXA | Total Hip Arthroplasty - Intravenous TXA | Total Knee Arthroplasty - Oral TXA | Total Knee Arthroplasty - Intravenous TXA | Total
Number analyzed (Participants) | 98 | 98 | 93 | 98 | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.84 (9.14) | 65.12 (7.32) | 66 (7.57) | 65.89 (7.28) | 65.2 (7.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 42 | 56 | 56 | 209
  Male | 43 | 56 | 37 | 42 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 8 | 9 | 31
  Not Hispanic or Latino | 90 | 92 | 85 | 89 | 356
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 5 | 7 | 6 | 21
  White | 92 | 87 | 75 | 81 | 335
  More than one race | 0 | 1 | 0 | 2 | 3
  Unknown or Not Reported | 3 | 5 | 7 | 7 | 22
Region of Enrollment [Number; unit: participants]
  United States | 98 | 98 | 93 | 98 | 387
American Society of Anesthesiology Status [Count of Participants; unit: Participants]
  ASA Level I | 3 | 5 | 3 | 2 | 13
  ASA Level II | 82 | 86 | 76 | 84 | 328
  ASA Level III | 13 | 7 | 14 | 11 | 45
  Unknown - ASA level missing | 0 | 0 | 0 | 1 | 1
Body Mass Index, kg/m^2 Mean (Standard Deviation) Unit of measure: Kg/m^2 [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (5.1) | 29.6 (4.3) | 29.4 (4.38) | 30.8 (5.1) | 29.62 (4.74)

OUTCOME MEASURES:

1. Primary Outcome: Calculated Blood Loss
Description: Calculated Blood loss (CBL) measured in mL, measured at baseline (before surgery) and in the post-operative care unit (after surgery). The following formula was used CBL = BV × (HctPre - HctPost), where BV = (k1 × H3) + (k2 × W) + k3. The variables for the formula are as followed:
  CBL: Calculated blood loss BV: Blood volume at baseline HctPre: Haematocrit before surgery HctPost: Haematocrit after surgery H: Patient height in meters W: Patient weight in kilograms
  Although measured at two time points (before and after surgery), the calculated value from those two time points is average across all participants and reported.
Time Frame: post-operative day 0
Measure: Mean (Standard Deviation); unit: CBL (ml)
Groups:
- Oral Tranexamic Acid (TXA) Total Hip Arthroplasty: 100 Total Hip Arthroplasty (THA) patients will be randomized to receive 1950 mg of oral TXA in the pre-operative area.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty: 100 Total Hip Arthroplasty (THA) patients will be randomized to receive 1 g of intravenous (IV) TXA upon transfer to the operating room.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Oral Tranexamic Acid (TXA) Total Knee Arthroplasty: 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1950 mg of oral TXA in the pre-operative area.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
- Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty: 100 Total Knee Arthroplasty (TKA) patients will be randomized to receive 1 g of intravenous (IV) TXA upon transfer to the operating room.
  Tranexamic Acid: Tranexamic acid (TXA) is an antifibrinolytic medication used to reduce bleeding in a variety of medical settings. Patients will be randomized to receive either oral or intravenous tranexamic acid.
Arm/Group | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty
Number analyzed (Participants) | 89 | 90 | 90 | 94
CBL (ml) | 842 (328) | 860 (313) | 799 (334) | 878 (348)

2. Secondary Outcome: Transfusion During Hospital Stay
Description: To assess how many participants required a blood transfusion during their hospital stay. This will be measured in binary responses (yes/no).
Time Frame: From Post-Operative Day 0 to Post-Operative Day 2
Measure: Number; unit: participants
Arm/Group | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty
Number analyzed (Participants) | 89 | 90 | 90 | 96
participants | 0 | 0 | 0 | 1

3. Secondary Outcome: Time to Discharge From Physical Therapy
Description: Time to discharge from physical therapy (in minutes)
Time Frame: From 48-72 hours after surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty
Number analyzed (Participants) | 87 | 87 | 89 | 92
minutes | 2091.33 (1203.17) | 1914.45 (1055.47) | 2244.55 (1327.44) | 2285.09 (1499.37)

4. Secondary Outcome: Length of Stay
Description: Hospital length of stay (in minutes)
Time Frame: After surgery to the time discharged from hospital (estimated 48-72 hours after surgery)
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty
Number analyzed (Participants) | 98 | 98 | 93 | 97
minutes | 2551.89 (1554.4) | 2138.6 (1126.71) | 2692.98 (1508.65) | 2852.55 (1511.05)

ADVERSE EVENTS:
Time Frame: From enrollment through study completion, an average of 1 week
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
  Adverse serious events were assessed over the course of the patient's participation in the research study.
Arm/Group | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty
All-Cause Mortality (participants affected / at risk) | 0/89 | 0/90 | 0/90 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/89 | 1/90 | 0/90 | 0/96
Other Adverse Events (participants affected / at risk) | 5/89 | 2/90 | 0/90 | 2/96
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty (N=89) | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty (N=90) | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty (N=90) | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty (N=96)
CVA, cerebrovascular accident (Vascular disorders) | 0 | 1 | 0 | 0 — New onset right hand numbness and weakness at 4 days postoperatively. Diagnosed with a stroke at the emergency room and started on Clopidrogrel.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Tranexamic Acid (TXA) Total Hip Arthroplasty (N=89) | Intravenous (IV) Tranexamic Acid (TXA) Total Hip Arthroplasty (N=90) | Oral Tranexamic Acid (TXA) Total Knee Arthroplasty (N=90) | Intravenous (IV) Tranexamic Acid (TXA) Total Knee Arthroplasty (N=96)
Complications (Blood and lymphatic system disorders) | 5 | 2 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-08): https://cdn.clinicaltrials.gov/large-docs/65/NCT04089865/Prot_SAP_000.pdf